CLINICAL TRIAL: NCT06300346
Title: Comparison Between Propofol, Ondansetron and Pregabalin for Control of Emetic Attacks During Caesarean Delivery With Spinal Anesthesia: Randomized Clinical Trial
Brief Title: Comparison Between Drugs for Control of Emetic Attacks During Caesarean Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ebtehal Ahmed Abdellattif, resident at Anesthesiology, Surgical Intensive Care and Pain Medicine department, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Soh-Med-23-12-02MS
Record Dates: First submitted 2024-02-14; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Emetic Attacks During Caesarean Delivery With Spinal Anesthesia
MeSH Terms: interventions — Propofol; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propofol (Active Comparator): 30 Patients will receive propofol as equal volumes of both 1% of propofol 10mg/ml and0.9% normal saline will be drawn in a 20-ml syringe before spinal puncture.
  Interventions: Drug: Propofol
- pregabalin (Active Comparator): 30 Patients will receive three capsules of pregabalin 100 mg once one hour before the surgical incision.
  Interventions: Drug: Propofol
- ondansetron (Active Comparator): 30 Patients will receive 4 mg ondansetron in 10 ml saline intravenously 5 min before spinal puncture.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Ondansetron
  Other Names: Pregabalin

SUMMARY:
Single shot spinal anesthesia is widely used for most surgical operations especially in obstetric such as hysterectomy, tubal ligation after vaginal delivery, cesarean and curettage etc.; however, in general, cesarean is considered as the most common indication for spinal anesthesia in pregnant women Intra-operative nausea and vomiting/retching (NVR) may be experienced by 20% to 80% of women undergoing cesarean section (CS) with subarachnoid anesthesia (SA) in the absence of antiemetic prophylaxis.

Different treatment options are available to reduce post operative nausea and vomiting (PONV) so we will make a Comparison between Propofol, Ondansetron and Pregabalin for Control of Emetic Attacks during Caesarean Delivery with Spinal Anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Age: 21-40 years old.
* Physical status American Society of Anesthesiologists (ASA)I&II.
* Body mass index (BMI) < 35&>20 kg/m2.
* Elective uncomplicated cesarean section under spinal anesthesia.

Exclusion Criteria:

* Patient refusal.
* Patients with known history of allergy to study drugs.
* Advanced hepatic, renal and respiratory diseases.
* Psychological and mental disorders.
* Patient with reduced level of consciousness.
* Hypertensive, cardiac, and diabetic patients.
* Patients receiving anticoagulants therapy or suspected coagulopathy.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-18 (Estimated); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of nausea and vomiting with spinal anesthesia | 5 months
  To compare between Propofol, Ondansetron and Pregabalin for control of emetic attacks during caesarean delivery with spinal anesthesia.

SECONDARY OUTCOMES:
Measurement of hemodynamics postoperative | 5 months
  Measurement of hemodynamics postoperative and Incidence of other side effects as :hypotension measured by non invasive blood pressure monitoring

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hirmanpour A, Safavi M, Honarmand A, Hosseini AZ, Sepehrian M. The comparative study of intravenous Ondansetron and sub-hypnotic Propofol dose in control and treatment of intrathecal Sufentanil-induced pruritus in elective caesarean surgery. J Res Pharm Pract. 2015 Apr-Jun;4(2):57-63. doi: 10.4103/2279-042X.155751. PMID 25984542
- [Background] Mokini Z, Genocchio V, Forget P, Petrini F. Metoclopramide and Propofol to Prevent Nausea and Vomiting during Cesarean Section under Spinal Anesthesia: A Randomized, Placebo-Controlled, Double-Blind Trial. J Clin Med. 2021 Dec 26;11(1):110. doi: 10.3390/jcm11010110. PMID 35011852
- [Background] Athavale A, Athavale T, Roberts DM. Antiemetic drugs: what to prescribe and when. Aust Prescr. 2020 Apr;43(2):49-56. doi: 10.18773/austprescr.2020.011. Epub 2020 Apr 1. PMID 32346211
- [Background] Elvir-Lazo OL, White PF, Yumul R, Cruz Eng H. Management strategies for the treatment and prevention of postoperative/postdischarge nausea and vomiting: an updated review. F1000Res. 2020 Aug 13;9:F1000 Faculty Rev-983. doi: 10.12688/f1000research.21832.1. eCollection 2020. PMID 32913634